CLINICAL TRIAL: NCT05582109
Title: A Single-arm, Open-label, Prospective, Phase II Clinical Study of Envafolimab, Lenvatinib Combined With TACE in the Treatment of Unresectable Locally Advanced Hepatocellular Carcinoma
Brief Title: Envafolimab, Lenvatinib Combined With TACE in the Treatment of Unresectable Locally Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-2022-0026
Record Dates: First submitted 2022-09-30; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-09

CONDITIONS: Objective Response Rate (ORR)
MeSH Terms: interventions — envafolimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab, Lenvatinib Combined With TACE (Experimental): Envafolimab, Lenvatinib Combined With TACE
  Interventions: Drug: Envafolimab, Lenvatinib Combined With TACE

INTERVENTIONS:
Drug: Envafolimab, Lenvatinib Combined With TACE — PD-L1 inhibitor

SUMMARY:
TACE lays a theoretical foundation for synergistic enhancement in combination with PD-1/PD-L1 immunosuppressive agents by reducing tumor burden and peripheral blood treg, improving the immune status of patients, reducing immune tolerance, and enhancing anti-tumor effects. TACE then causes locally treated tumor cell death and releases tumor-specific antigens, which further induce tumor-associated antigen-specific responses due to this immunogenic cell death (ICD), thereby activating the immune system to attack tumor cells.

This is a single-arm, open-label, exploratory clinical study to evaluate the efficacy and safety of Envafolimab, Lenvatinib combined with TACE in the treatment of unresectable locally advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent before enrollment;
2. Age > 18, both male and female;
3. Pathologically confirmed unresectable locally advanced hepatocellular carcinoma;
4. With measurable lesions (according to RECIST 1.1 criteria, non-lymph node lesions CT scan long diameter ≥ 10 mm, lymph node lesions CT scan short diameter ≥ 15 mm);
5. ECOG PS: 0 to 1;
6. Expected survival greater than 12 weeks;
7. Vital organ function in accordance with the following requirements (excluding any blood components and cell growth factors within 14 days): 1) blood routine: neutrophils ≥ 1.5 × 10^9/L platelet count ≥ 100 × 10^9/L hemoglobin ≥ 90 g/L; 2) liver and kidney function: serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula); total bilirubin (TBIL) ≤ 1.5 times ULN; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤ 2.5 ULN (≤ 5ULN if liver function abnormalities are due to liver metastases); urine protein < 2 +; if urine protein ≥ 2 +,24-hour urine protein must show protein ≤ 1g;
8. Normal coagulation, no active bleeding and thrombosis disease 1) international normalized ratio INR ≤ 1.5 × ULN; 2) partial thromboplastin time APTT ≤ 1.5 × ULN; 3) prothrombin time PT ≤ 1.5 × ULN;
9. Non-surgically sterilized or female patients of childbearing age who need to use a medically recognized contraceptive (such as an intrauterine device, contraceptive pills or condom) during study treatment and within 3 months after the end of study treatment; non-surgically sterilized female patients of childbearing age must have a negative serum or urine HCG test within 7 days before study enrollment; and must be non-lactating; non-surgically sterilized or male patients of childbearing age who need to agree to use a medically recognized contraceptive during study treatment and within 3 months after the end of study treatment with their spouses.
10. The subject voluntarily joined this study with good compliance and cooperation in safety and survival follow-up.

Exclusion Criteria:

1. The subject has previous or concurrent other malignant tumors (except cured cutaneous basal cell carcinoma and cervical carcinoma in situ);
2. Previous treatment with other PD-1/PD-L1 inhibitors can not be enrolled; known that the subject has previous hypersensitivity to macromolecular protein preparations, or known to the applied drug components;
3. The subject has any active autoimmune disease or history of autoimmune diseases (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, previous thyroid surgery can not be included; the subject has vitiligo or has complete remission of asthma in childhood, adults do not need any intervention can be included; the subject requires bronchodilators for medical intervention of asthma can not be included);
4. The subject is using immunosuppressive agents, or systemic, or absorbable local hormone therapy to achieve immunosuppressive purposes (dose > 10 mg/day prednisone or other effective hormones), And continue to use within 2 weeks before enrollment;
5. Ascites or pleural effusion with clinical symptoms, requiring therapeutic puncture or drainage;
6. Cardiac clinical symptoms or diseases that are not well controlled,For example: (1) NYHA class A2 or higher heart failure; (2) unstable angina pectoris; (3) myocardial infarction within 1 year; (4) patients with clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention;
7. Subjects are still using traditional Chinese medicine immunomodulators within 2 weeks before enrollment;
8. Subjects have active infection or unexplained fever > 38.5 degrees during screening and before the first dose (subjects can be enrolled due to tumor-induced fever as judged by the investigator);
9. Patients with objective evidence of previous and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, and severely impaired pulmonary function;
10. Subjects with congenital or acquired immunodeficiency, such as HIV infection, or active hepatitis (transaminase does not meet the inclusion criteria, hepatitis B reference: HBV DNA ≥ 1000 IU/ml; hepatitis C reference: HCV RNA ≥ 1000 IU/ml); chronic hepatitis B virus carriers, HBV DNA < 2000 IU/ml, must receive concurrent antiviral therapy during the trial to be enrolled;
11. Live vaccines less than 4 weeks prior to study medication or likely during the study;
12. Subject has a known history of psychiatric drug abuse, alcoholism, or drug abuse;
13. The subject had received treatment with traditional Chinese medicine within 4 weeks before the first treatment;
14. The investigator considered that the subject should be excluded from this study, for example, the investigator judged that the subject had other factors that might cause forced halfway termination of this study, for example, other serious diseases (including mental illness) required concomitant treatment, there were serious laboratory abnormalities, accompanied by family or social factors, which would affect the safety of the subject, or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 36 month
  Refers to the proportion of patients who achieve a pre-specified reduction in tumor size and maintain the minimum time limit

SECONDARY OUTCOMES:
Overall survival | up to 36 month
  Time from randomization to death from any cause (for subjects who were lost to follow-up prior to death, the time of last follow-up was generally calculated as the time of death)
Progression Free Survival | up to 12 month
  Time to first occurrence of disease progression or death from any cause at randomization
Adverse Events | up to 36 month
  Any untoward medical occurrence in a patient or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment

IPD SHARING:
Plan to Share IPD: Undecided